CLINICAL TRIAL: NCT02869997
Title: Evaluation of the Prognostic Value of the Suppression Ratio Evaluated by BIS Among Patients Admitted to the ICU for Cardiac Arrest
Acronym: SACRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P/2012/128
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): arm wherein all patients Suppression Ratio evaluated by BIS will be collected
  Interventions: Device: Aspect BIS XP (A-2000) Bispectral Index Patient Monitor

INTERVENTIONS:
Device: Aspect BIS XP (A-2000) Bispectral Index Patient Monitor

SUMMARY:
The aim of this study is to evaluate the prognostic value of the suppression ratio monitored by Bispectral Index for prediction of neurologic outcome after cardiac arrest. All patient admitted to our intensive care unit after a cardiac arrest are included. The results of the suppression ratio will be collected in the 6 first hours of admission. We will evaluate the link between suppression ratio and cerebral performance category score collected at three months.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Cardiac arrest admitted to the ICU

Exclusion Criteria:

- Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-08; Primary Completion 2014-09 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Cerebral Performance Category score | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: François Belon, MD, Principal Investigator — CHRU Besançon
Locations (1):
- CHRU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No